CLINICAL TRIAL: NCT00244270
Title: Cystic Fibrosis and Totally Implantable Vascular Access Devices: Evaluation of the Incidence of Venous Thrombosis Related to the Catheter and Study of the Genetic and Acquired Risk Factors
Brief Title: Cystic Fibrosis and Totally Implantable Vascular Access Devices
Acronym: RITHM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P041202
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis; Venous Thrombosis
Keywords: totally implantable vascular access devices; thromboembolism; genetic susceptibility to venous thrombosis.
MeSH Terms: conditions — Cystic Fibrosis; Venous Thrombosis; Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): totally implantable vascular access device
  Interventions: Device: totally implantable vascular access device

INTERVENTIONS:
Device: totally implantable vascular access device — totally implantable vascular access device

SUMMARY:
The purpose of this study is to evaluate the incidence of venous thrombosis occurring on totally implantable vascular access devices in cystic fibrosis patients who need a new device (it can be the first one or a subsequent one) and to study the genetic risk factors of thrombosis adjusted to the acquired ones.

It is a nationwide cohort study planned for two years with a six month follow up period. The expected number of inclusion is 50 patients each year, that is to say 100 for the whole study.

In cystic fibrosis, pulmonary exacerbations necessitate repeated intravenous antibiotics, but the peripheral blood accesses become precarious with time, leading to the indication of a central venous device. It is important to take a lot of precautions to protect vascular access. This allows the patient to have a dramatic improvement in life expectancy with such life-long devices (ONM, French National Observatory France 2003 : median at 36 years). Venous thrombosis can cause a superior cava syndrome, a pleural effusion or a pulmonary embolism. The risk of thrombosis is significant; retrospectively, it has been evaluated to be between 4 and 16% in the publications. This rate may be higher due to the fact that venous thrombosis may remain asymptomatic, and therefore silent, but they lead to the same risk of vascular access loss.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the incidence of venous thrombosis occurring on totally implantable vascular access devices in cystic fibrosis patients who need a new device (it can be the first one or a subsequent one) and to study the genetic risk factors of thrombosis adjusted to the acquired ones.

It is a nationwide cohort study planned for two years with a six month follow up period. The expected number of inclusion is 50 patients each year, that is to say 100 for the whole study.

In cystic fibrosis, pulmonary exacerbations necessitate repeated intravenous antibiotics, but the peripheral blood accesses become precarious with time, leading to the indication of a central venous device. It is important to take a lot of precautions to protect vascular access. This allows the patient to have a dramatic improvement in life expectancy with such life-long devices (ONM, French National Observatory France 2003 : median at 36 years). Venous thrombosis can cause a superior cava syndrome, a pleural effusion or a pulmonary embolism. The risk of thrombosis is significant; retrospectively, it has been evaluated to be between 4 and 16% in the publications. This rate may be higher due to the fact that venous thrombosis may remain asymptomatic, and therefore silent, but they lead to the same risk of vascular access loss.

This prospective study will try to identify venous thrombosis whatever they are - symptomatic or silent - and to identify the genetic and acquired risk factors, the circumstances of occurrence and the current therapeutic modalities. Furthermore, the setting up of an early treatment on still asymptomatic thrombosis allows the researchers to hope for a prompt resolution of the thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Children or adults with cystic fibrosis (identified either by 2 abnormal sweat tests and/or two CFTR [cystic fibrosis transmembrane conductance regulator] mutations) who need a totally implantable vascular access device.
* Signed informed consent

Exclusion Criteria:

* Refusal of participation in the study
* Patients on a waiting list for pulmonary or hepatic transplantation
* Patients who received a pulmonary or hepatic graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2005-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
There is no primary outcome measure specified for this study. | during de study
  There is no primary outcome measure specified for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Munck, MD, Principal Investigator — Hôpital Robert Debré, APHP, France